CLINICAL TRIAL: NCT01745185
Title: Immune Response in Subjects With Fabry Disease Who Are Switching From Agalsidase Alfa to Agalsidase Beta
Status: Completed | Type: Observational
Sponsor: O & O Alpan LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 12-CFCT-03
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; immunity; antibody
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fabry disease switch group: Subjects will include individuals with Fabry disease who are switching from agalsidase alfa to agalsidase beta
- Control Group: Controls will include individuals with Fabry disease who have only received agalsidase beta as treatment in their lifetime.

SUMMARY:
This study is a prospective active comparator study to assess the immune response elicited by human recombinant agalsidase therapy in subjects who are switching from agalsidase alfa to agalsidase beta with Fabry disease. Fabry disease is an X-linked lysosomal storage disorder, due to deficient alpha-galactosidase A activity. The progressive accumulation of globotriaosylceramide (GL-3) in the lysosomes of the vascular endothelial cells of multiple organ systems like the kidneys, heart, skin, and brain, leads to a microvascular disease. In Fabry disease, nephropathy dominates and renal function impairment occurs as a result of accumulation of GL-3 in renal cells

DETAILED DESCRIPTION:
Clinically, the development of an immune response is anticipated in a number of patients treated with any recombinant human proteins and suggested to be more common especially when the native protein is deficient or absent as many male patients with Fabry disease.

The immune response that results in the development of antibodies against the infused proteins may affect the clinical outcome of enzyme replacement therapy by the development of hypersensitivity, anaphylactoid, or febrile reactions, or may lead to the development of cytokine release and a generalized inflammatory response or immune complex formation. Furthermore, the mounted immune response may lead to inactivation or degradation of the recombinant enzyme or may change the pharmacokinetic and pharmacodynamic properties of the therapeutic protein.

The different rates of antibody formation with agalsidase alfa and agalsidases beta are often attributed to differences in techniques used to measure antibody formation. However, other factors such as host, structural similarity of the infused protein and tertiary structural difference such as glycosylation may lead to differences in the immune response. Among the factors that may affect host response are also the dose and the infusion frequency. Although agalsidase alfa and beta are derived from the same complementary DNA sequence there are minor differences in glycosylation patterns, and different dosing is used, 0.2 mg per kg every other week for agalsidase alfa, 1.0 mg per kg for agalsidase beta.

The investigator hypothesize that although the observation that the antibodies exhibit in vitro neutralizing capacity may suggest the presence of a single immunogenic epitope for both human recombinant alpha-galactosidases, the immunogenicity may not be similar for both agalsidase alfa and beta, and thus the differences in immune response will be determined by the host factors and the escalating dose of infused protein.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Fabry disease
* Have been treated with ERT using recombinant human agalsidase A.

Exclusion Criteria:

* If the diagnosis of Fabry disease is not confirmed
* If the subject or guardian is not able to provide consent
* Any chronic immunosuppressive state or therapy such as patients on dialysis or post-transplantation immunosuppressive therapy.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 30 subjects of (7 and above) who meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2015-04-07 (Actual); Study Completion 2016-08-07 (Actual)

PRIMARY OUTCOMES:
Monitoring antibody formation against agalsidase alfa and beta | 12 months
  Blood samples will be collected prior to infusion (screening & month 12). At baseline, antibodies against agalsidase alfa and beta measured, and at 12 months, antibodies against agalsidase beta will be measured by ELISA technique and will be isotyped immunoglobulins (IgG, IgA, IgM, or IgE). Positive samples will subsequently tested for enzyme neutralizing activity using an in vitro assay. Antibody measurements will be done by Shire Human Genetics Therapies, INC.

SECONDARY OUTCOMES:
Measurement of plasma/urine Gb3 and plasma lyso-Gb3 | 12 months
  Plasma samples collected after at least 8 hours of fasting prior to the blood draw. Plasma and urine samples (Gb3 only) analyzed using mass spectrometry. Gb3 measurements will be performed by Shire HGT.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Goker-Alpan, MD, Principal Investigator — O & O Alpan LLC
Locations (1):
- O&O Alpan, Fairfax, Virginia, United States

REFERENCES:
- [Background] Benichou B, Goyal S, Sung C, Norfleet AM, O'Brien F. A retrospective analysis of the potential impact of IgG antibodies to agalsidase beta on efficacy during enzyme replacement therapy for Fabry disease. Mol Genet Metab. 2009 Jan;96(1):4-12. doi: 10.1016/j.ymgme.2008.10.004. Epub 2008 Nov 20. PMID 19022694